CLINICAL TRIAL: NCT05878990
Title: Quit & Fit 2.0: Feasibility and Usability Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2022-0894
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Smoking Cessation
Keywords: smoking; smoking cessation; smoking behavior; culturally tailored tobacco cessation intervention
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally-tailored Tobacco Treatment Intervention (Active Comparator): Upon consent, participants will complete a baseline survey, receive the home Carbon monoxide monitor and instructions on how to use, and be scheduled for weekly telephone calls with a certified tobacco treatment specialist (CTTS) for 6 weeks. The culturally-tailored tobacco intervention content by week via telephone call with the CTTS includes among others: Reasons and Motivations for Quitting, Benefits of Quitting, Stress Management and Discussion about Environmental Influences. Participants will also receive weekly Culturally-tailored Content Newsletters emailed after their weekly cessation counseling session.
  Interventions: Behavioral: Culturally-tailored Tobacco Treatment; Behavioral: Culturally-tailored Content Newsletters
- Preference-Driven Culturally-tailored Tobacco Treatment Intervention (Active Comparator): Upon consent, participants will complete a baseline survey, receive the home Carbon monoxide monitor and instructions on how to use, and be scheduled for weekly telephone calls with a certified tobacco treatment specialist (CTTS) for 6 weeks. The culturally-tailored tobacco intervention content by week via telephone call with the CTTS includes among others: Reasons and Motivations for Quitting, Benefits of Quitting, Stress Management and Discussion about Environmental Influences. Participants will complete the one-item Control Preference Scale and receive either an Active Content Newsletter or Passive Content Newsletter emailed after their weekly cessation counseling session.
  Interventions: Behavioral: Culturally-tailored Tobacco Treatment; Behavioral: Control Preference Scale; Behavioral: Active Content Newsletter or Passive Content Newsletter

INTERVENTIONS:
Behavioral: Culturally-tailored Tobacco Treatment — Weekly telephone calls with a certified tobacco treatment specialist (CTTS) for 6 weeks. The culturally-tailored tobacco intervention content by week via telephone call with the CTTS includes among others: Reasons and Motivations for Quitting, Benefits of Quitting, Stress Management and Discussion about Environmental Influences.
Behavioral: Culturally-tailored Content Newsletters — Weekly newsletters covering topics such as Race and Smoking, Nicotine Replacement Therapy (NRT) Reasons and Motivations for Quitting, Benefits of Quitting and other related topics.
  Arms: Culturally-tailored Tobacco Treatment Intervention
Behavioral: Control Preference Scale — Survey to elicit preference on the decision-making interaction with healthcare provider. The survey uses a 5 point scale from 1 to 5 with 1 or 2 points representing Active Control Preference; 3 or 4 representing a Collaborative Control Preference and 5 representing a Passive Control Preference.
  Arms: Preference-Driven Culturally-tailored Tobacco Treatment Intervention
Behavioral: Active Content Newsletter or Passive Content Newsletter — Based on the answers to the Control Preference Scale, participants will receive the appropriate weekly newsletter (active content or passive content). Newsletters are covering topics such as Race and Smoking, Nicotine Replacement Therapy (NRT) Reasons and Motivations for Quitting, Benefits of Quitting and other related topics presented in a more passive or active manner.
  Arms: Preference-Driven Culturally-tailored Tobacco Treatment Intervention

SUMMARY:
Pilot randomized controlled trial to compare tobacco cessation rates of two arms: a 6-week culturally tailored tobacco cessation intervention versus a 6-week personalized culturally-tailored tobacco cessation intervention among African American women.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as an African American woman
* Currently smoke 5 cigarettes per day or more
* Has smoked daily for the past one year
* Able to provide informed consent
* Generally good health as determined by medical history

Exclusion Criteria:

* Currently pregnant
* Diagnosis of cardiovascular disease
* Diagnosis of lung disease
* Diagnosis of mental illness
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as an African American woman
Enrollment: 22 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carter-Bawa, PhD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Meridian Health - Center for Discovery and Innovation, Nutley, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Ries LAG, Melbert D, Krapcho M. SEER cancer statistics review, 1975-2005. 2008. 2. American Cancer Society. Cancer facts and figures for African Americans: 2022. 3. Siegel R, Naishadham D, Jemal A. Cancer statistics, 2021. CA Cancer J Clin. 2021;62(1):10-29. 4. Singh GK, Williams SD, Siahpush M, Mulhollen A. Socioeconomic, rural-urban, and racial inequalities in US cancer mortality: Part I-all cancers and lung cancer and part II-colorectal, prostate, breast, and cervical cancers. J Cancer Epidemiol. 2011;2011:107497. 5. Haiman CA, Stram DO, Wilkens LR, et al. Ethnic and racial differences in the smoking-related risk of lung cancer. N Engl J Med. 2006;354(4):333-342. 6. Wang Y, Beydoun MA. The obesity epidemic in the united states--gender, age, socioeconomic, racial/ethnic, and geographic characteristics: A systematic review and meta-regression analysis. Epidemiol Rev. 2007;29:6-28. 7. Roger VL, Go AS, Lloyd-Jones DM, et al. Heart disease and stroke statistics--2012 update: A report from the american heart association. Circulation. 2012;125(1):e2-e220.
- [Background] 8. Dubowitz T, Heron M, Bird CE, et al. Neighborhood socioeconomic status and fruit and vegetable intake among whites, blacks, and mexican americans in the united states. Am J Clin Nutr. 2008;87(6):1883-1891. 9. U.S. physical activity statistics: 2007 state demographic data comparison. 2008. 10. Marshall SJ, Jones DA, Ainsworth BE, Reis JP, Levy SS, Macera CA. Race/ethnicity, social class, and leisure-time physical inactivity. Med Sci Sports Exerc. 2007;39(1):44-51. 11. Bassuk SS, Manson JE. Physical activity and cardiovascular disease prevention in women: A review of the epidemiologic evidence. Nutr Metab Cardiovasc Dis. 2010;20(6):467-473. 12. Glasgow RE, Lichtenstein E, Marcus AC. Why don't we see more translation of health promotion research to practice? rethinking the efficacy-to-effectiveness transition. Am J Public Health. 2003;93(8):1261-1267. 13. Swan GE, Ward MM, Carmelli D, Jack LM. Differential rates of relapse in subgroups of male and female smokers. J Clin Epidemiol. 1993;46(9):1041-1053. 14. Pirie PL, Murray DM, Luepker RV. Gender differences in cigarette smoking and quitting in a cohort of young adults. Am J Public Health. 1991;81(3):324-327. 15. Pomerleau CS, Zucker AN, Namenek Brouwer RJ, Pomerleau OF, Stewart AJ. Race differences in weight concerns among women smokers: Results from two independent samples. Addict Behav. 2001;26(5):651-663.
- [Background] 16. Berg CJ, Thomas JL, An LC, et al. Change in smoking, diet, and walking for exercise in blacks. Health Educ Behav. 2012;39(2):191-197. 17. Ussher MH, Taylor AH, Faulkner GE. Exercise interventions for smoking cessation. Cochrane Database Syst Rev. 2014;8:CD002295. 18. Marcus BH, Albrecht AE, Niaura RS, Abrams DB, Thompson PD. Usefulness of physical exercise for maintaining smoking cessation in women. Am J Cardiol. 1991;68(4):406-407. 19. Marcus BH, King TK, Albrecht AE, Parisi AF, Abrams DB. Rationale, design, and baseline data for commit to quit: An exercise efficacy trial for smoking cessation among women. Prev Med. 1997;26(4):586-597. 20. Marcus BH, Albrecht AE, King TK, et al. The efficacy of exercise as an aid for smoking cessation in women: A randomized controlled trial. Arch Intern Med. 1999;159(11):1229-1234. 21. Marcus BH, Albrecht AE, Niaura RS, et al. Exercise enhances the maintenance of smoking cessation in women. Addict Behav. 1995;20(1):87-92. doi: 0306460394000484 [pii]. 22. Marcus BH, Lewis BA, King TK, et al. Rationale, design, and baseline data for commit to quit II: An evaluation of the efficacy of moderate-intensity physical activity as an aid to smoking cessation in women. Prev Med. 2003;36(4):479-492. 23. Whiteley JA, Napolitano MA, Lewis BA, et al. Commit to quit in the YMCAs: Translating an evidence-based quit smoking program for women into a community setting. Nicotine Tob Res. 2007;9(11):1227-1235.
- [Background] 24. Webb MS, Baker EA, Rodriguez de Ybarra D. Effects of culturally specific cessation messages on theoretical antecedents of behavior among low-income african american smokers. Psychol Addict Behav. 2010;24(2):333-341. 25. Travier N, Agudo A, May AM, et al. Longitudinal changes in weight in relation to smoking cessation in participants of the EPIC-PANACEA study. Prev Med. 2012;54(3-4):183-192. 26. Filozof C, Fernandez Pinilla MC, Fernandez-Cruz A. Smoking cessation and weight gain. Obes Rev. 2004;5(2):95-103. 27. Grunberg NE. A neurobiological basis for nicotine withdrawal. Proc Natl Acad Sci U S A. 2007;104(46):17901-17902. 28. Mineur YS, Abizaid A, Rao Y, et al. Nicotine decreases food intake through activation of POMC neurons. Science. 2011;332(6035):1330-1332. 29. Seeley RJ, Sandoval DA. Neuroscience: Weight loss through smoking. Nature. 2011;475(7355):176-177. 30. Whittaker R, McRobbie H, Bullen C, Borland R, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2012;11:CD006611. 31. Stead LF, Perera R, Lancaster T. Telephone counselling for smoking cessation. Cochrane Database Syst Rev. 2006;(3)(3):CD002850. 32. Mottillo S, Filion KB, Belisle P, et al. Behavioural interventions for smoking cessation: A meta-analysis of randomized controlled trials. Eur Heart J. 2009;30(6):718-730. 33. Migneault JP, Dedier JJ, Wright JA, et al. A culturally adapted telecommunication system to improve physical activity, diet quality, and medication adherence among hypertensive african-americans: A randomized controlled trial. Ann Behav Med. 2012;43(1):62-73. 34. Mobile technology fact sheet. http://www.pewinternet.org/fact-sheets/mobile-technology-fact-sheet/. Updated January 2014.
- [Derived] Carter-Bawa L, Binstock J, Vielma AG, Shoulders EN, Adams-Campbell L. EmpowerHer-a smoke-free future: a feasibility study examining the feasibility and acceptability of a culturally concordant tobacco treatment intervention in African American women. Pilot Feasibility Stud. 2025 May 31;11(1):75. doi: 10.1186/s40814-025-01664-y. PMID 40450357

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Culturally-tailored Tobacco Treatment Intervention
Started | 22
Completed | 14
Not Completed | 8
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Culturally-tailored Tobacco Treatment Intervention
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the 6-week Tobacco Treatment Intervention
Description: Examine the feasibility of a 6-week community-based culturally tailored tobacco treatment intervention to a preference driven culturally-tailored tobacco treatment intervention targeted to African American women by assessing the number of participants that complete all 6-week tobacco treatment calls.
Time Frame: Post intervention completion - At 6 weeks
Population: Participants who consented and initiated intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Culturally-tailored Tobacco Treatment Intervention
Number analyzed (Participants) | 22
Participants | 14

2. Primary Outcome: Accessibility and Satisfaction of the 6-week Tobacco Treatment Intervention
Description: Examine the acceptability and satisfaction of a 6-week community-based culturally-tailored tobacco treatment intervention to a preference driven culturally-tailored tobacco treatment intervention targeted to African American women using the 17-item Acceptability & Satisfaction Questionnaire. Accessibility and Satisfaction and measured using a score that ranges from 17 to 68 with higher scores representing higher Accessibility and Satisfaction.
Time Frame: Post intervention completion - At 6 weeks
Population: Participants who completed the intervention and the Accessibility and Satisfaction questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Culturally-tailored Tobacco Treatment Intervention
Number analyzed (Participants) | 14
score on a scale | 56.08 (5.14)

3. Secondary Outcome: Effectiveness of the Intervention (Fagerstrom Test)
Description: Evaluate the effectiveness of a 6-week community-based culturally-tailored tobacco treatment intervention using the Fagerstrom Test for Nicotine Dependence. The Fagerström Test for Nicotine Dependence is a psychometrically-validated self-report 6-item tool to measure an individuals' level of nicotine dependence with a total scale score ranging from 0-10 with higher scores indicative of higher levels of nicotine dependence.
Time Frame: Post intervention completion - At 6 weeks
Population: Participants who completed the Fagerström Test for Nicotine Dependence after completing the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Culturally-tailored Tobacco Treatment Intervention
Number analyzed (Participants) | 14
score on a scale | 2.5 (2.07)

4. Secondary Outcome: Effectiveness of the Intervention (Expired Air Carbon Monoxide Readings)
Description: Evaluate the effectiveness of a 6-week community-based culturally-tailored tobacco treatment intervention using expired air carbon monoxide readings. Higher carbon monoxide readings are associated with worse outcomes.
Time Frame: 6 weeks post intervention
Population: Participants who completed the air carbon monoxide readings after completing the intervention.
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Culturally-tailored Tobacco Treatment Intervention
Number analyzed (Participants) | 14
ppm | 7.125 (3.72)

5. Secondary Outcome: Effectiveness of Intervention
Description: Evaluate the effectiveness of a 6-week community-based culturally-tailored tobacco treatment intervention using Stage of Change for Tobacco Cessation. The "Stage of Change for Tobacco Cessation" measures participants intention to quit smoking and has 4 categories: No Plans to Quit / Within the Next 6 Months/ Within the Next 30 Days / Quit. Results were compared to baseline Stage of Change.
Time Frame: 6 weeks post intervention
Population: Baseline and post intervention Stage of Change
Measure: Count of Participants; unit: Participants
Groups:
- Culturally-tailored Tobacco Treatment Intervention: Baseline Stage of Change
- Culturally-tailored Tobacco Treatment Intervention - Post Intervention: Post intervention Stage of Change
Arm/Group | Culturally-tailored Tobacco Treatment Intervention | Culturally-tailored Tobacco Treatment Intervention - Post Intervention
Number analyzed (Participants) | 14 | 14
Participants
  No Plans to Quit | 0 | 0
  Within the Next 6 Months | 5 | 5
  Within the Next 30 Days | 9 | 6
  Quit | 0 | 3

ADVERSE EVENTS:
Time Frame: 6 weeks of intervention
Arm/Group | Culturally-tailored Tobacco Treatment Intervention
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
A decision was made not to randomize participants since the focus of the study was the feasibility of the intervention. Therefore, there was never a second cohort of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT05878990/Prot_SAP_000.pdf